CLINICAL TRIAL: NCT06523777
Title: Optimizing Prostate Cancer Care: Integrating Risks, Benefits and Patient Experiences in the New Era of Molecular Imaging
Brief Title: PRISM: Patient Experiences With PET Imaging in Prostate Cancer
Acronym: PRISM
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000037284; 1R01CA281959-01 (NIH)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine patient experiences, health-related quality of life, and decision-making associated with PET imaging for prostate cancer. In particular, Prostate Specific Membrane Antigen (PSMA) PET, a new and more sensitive form of imaging that can help identify metastatic cancer earlier and more reliably.

DETAILED DESCRIPTION:
The primary objective is to measure health related quality of life among patients with prostate cancer who are undergoing prostate specific membrane positron emission tomography (PSMA-PET) imaging. This will be assessed in four domains: cancer related anxiety, decisional conflict, health related quality of life (physical functioning) and health preferences.

The secondary objective is to conduct longitudinal in-depth qualitative interviews to better explore patient experiences and perspectives on PET imaging.

Study Design Investigators will conduct a longitudinal explanatory sequential mixed methods study consisting of two phases. In the first phase, serial quantitative psychological (anxiety, uncertainty) and HRQoL survey data from patients undergoing PET imaging in routine clinical care will be collected. In the second phase, a subset of patients from phase 1 who have completed initial surveys will be recruited and conduct longitudinal in-depth qualitative interviews to better explore patient experiences and perspectives on PET imaging.

Patient clinical and sociodemographic data will be collected through automated extraction from the medical record (EPIC) into the REDcap database through collaboration with JDAT. For fields that are not populated via automated methods we will manually enter information via abstraction of the patient's medical record (EPIC).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of prostate cancer
* Scheduled for their FIRST PSMA PET scan for prostate cancer
* English-speaking
* Willing and able to complete 4 surveys electronically or on paper at 3 timepoints (within 1 month after PET scan, 3-6 months, 12 months)
* Able to use mobile device (smartphone or tablet) or computer with web access to complete study surveys or able to complete paper surveys

Exclusion Criteria:

* Lack of access to a mobile device (smartphone or tablet) or computer with web access or unable to receive surveys by mail.
* Unable to give consent and be enrolled
* PET scan is being conducted within a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with documented diagnosis of prostate cancer undergoing PSMA-PET imaging, including participants along the disease spectrum (all grades, stages, and indications for imaging). Participants will be identified and screened from all referrals to PET imaging and contacted by a study coordinator.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Memorial Anxiety Scale for Prostate Cancer (MAX-PC) | baseline, 3-6 months, and 12 months
  An 18-item instrument assessing frequency of anxiety in response to prostate cancer with 4 Likert responses ranging from 0 (not at all) to 3 (often); total score range 0 to 54). Higher scores indicate more anxiety.
Change in Decisional Conflict Scale (DCS) | baseline, 3-6 months, and 12 months
  A 16-item instrument using a 5-point Likert scale, ranging from 0 (strongly agree)-4 (strongly disagree), that has been widely applied to understand decision-making in prostate cancer. Higher scores indicate greater degrees of decisional conflict. DCS subscales include patient perceptions of uncertainty in choosing among treatment options, the contribution of modifiable factors (e.g., feeling uninformed), and effectiveness of decision-making (e.g., satisfaction with the choice). Total and subscale scores range from 0 to 100.
Change in Expanded Prostate Cancer Index Composite Short Form (EPIC-26) | baseline, 3-6 months, and 12 months
  A 26 item prostate cancer specific health-related quality of life (HRQOL) questionnaire assessing urinary incontinence, urinary irritative/obstructive, bowel, sexual and hormonal domains. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Change in EuroQol-5 Dimension (EQ-5D) | baseline, 3-6 months, and 12 months
  The instrument assesses five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. EQ-5D values can be converted to calculate health utilities that will be used for estimation of quality adjusted life years in decision analytic modeling. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions. A utility score was obtained by using a weighted combination of the levels of the five dimension-scales.

SECONDARY OUTCOMES:
Qualitative interviews on patient experiences and perspectives on PET imaging. | baseline, 3-6 months, and 12 months
  Longitudinal in-depth qualitative interviews to better explore patient experiences and perspectives on PET imaging to assess emergent themes. A subset of patients will be invited to participate in parallel in depth focused interviews occurring at three time points matching those of the surveys. Sample size will be dynamic and assessed based on emergent themes that become apparent during coding and analysis of interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leapman, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - Yale New Haven Health Bridgeport Hospital - Park Ave Medical Center, Bridgeport, Connecticut
  - Griffin Hospital, Derby, Connecticut
  - Yale New Haven Health Greenwich Hospital, Greenwich, Connecticut
  - Radiology and Biomedical Imaging - New Haven - Smilow Cancer Hospital (North Pavilion):, New Haven, Connecticut
  - Saint Raphael's Radiology and Biomedical Imaging, Basement Location., New Haven, Connecticut
  - Yale New Haven Health Lawrence & Memorial Hospital, New London, Connecticut
  - Yale New Haven Health Westerly Hospital, Westerly, Rhode Island

IPD SHARING:
Plan to Share IPD: No